CLINICAL TRIAL: NCT07393919
Title: Safe Discontinuation of Antidepressants in Individuals With Clinically Remitted Depressive Disorders
Brief Title: Discontination of Antidepressants in Remitted Depression
Acronym: DISCARD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other); Centro Ricerche Cliniche di Verona (Other)
Responsible Party: Principal Investigator, Giovanni Ostuzzi, Principal Investigator; Assistant Professor; MD; PhD, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSTUZZI_PRIN_PNRR2022_M4C2_INV; 2023-509377-23 (EudraCT Number)
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder
Keywords: depression; antidepressants; clinically remitted depressive disorder; discontinuation of the antidepressant
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Individuals will be randomized 1:1 to linear or hyperbolic tapering, The sequence of treatments will be randomly permuted in blocks of constant size. The allocation will be stratified by (a) recruiting centre; (b) individuals at high- vs. low-risk of withdrawal symptoms,
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor and the statistician will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Linear tapering (Active Comparator): Antidepressant (AD) dose will be reduced by fixed amounts (generally 50% of the minimum effective dose) every 2 weeks, according to pre-defined schedules, with the aim of reaching 50% of the minimum effective dose (as defined in the AIFA Summary of Product Characteristics), and finally discontinuing the AD after 4 to 10 weeks (depending on the initial dose). This approach is similar to the tapering schedules commonly used in current clinical practice. Any SSRI, SNRI, tricyclic antidepressant, and vortioxetine will be allowed.
  Interventions: Drug: Linear tapering
- Hyperbolic tapering (Active Comparator): Antidepressant (AD) dose will be reduced by 20-25% every 2 weeks, according to pre-defined schedules adapted from the Maudsley Hospital Guidelines (Taylor, 2021), with the aim of reaching at least 20% of the minimum effective dose (as defined in the AIFA Summary of Product Characteristics), and finally discontinuing the AD after 12 to 20 weeks (depending on the initial dose). Any SSRI, SNRI, tricyclic antidepressant, and vortioxetine will be allowed.
  Interventions: Drug: Hyperbolic tapering

INTERVENTIONS:
Drug: Hyperbolic tapering — The dose will be reduced by 20-25% every 2 weeks.
  Arms: Hyperbolic tapering
Drug: Linear tapering — Dose will be reduced by fixed amounts (generally 50% of the minimum effective dose) every 2 weeks.
  Arms: Linear tapering

SUMMARY:
Overprescribing and long-term use of antidepressants (ADs) are common and may increase the risk of adverse effects and withdrawal symptoms when discontinuation is attempted. Although several discontinuation strategies have been proposed, empirical evidence comparing different tapering approaches is limited. In particular, hyperbolic tapering has been suggested as a potentially safer and more effective alternative to standard linear tapering, but no randomized trials have directly compared these strategies.

This study is a pragmatic, multicentre, open-label, parallel-group, superiority randomized trial designed to compare two antidepressant discontinuation strategies-linear tapering and hyperbolic tapering-in adults with remitted depressive disorders. Eligible participants are adults aged 18 years or older with currently remitted depressive disorders who have been taking antidepressants for at least six months and are considered clinically appropriate candidates for discontinuation.

Participants will be recruited in outpatient psychiatric settings, with the involvement of general practitioners and other medical specialists. After baseline assessment, participants will be randomized to either a linear tapering strategy, consisting of dose reductions of 50% of the minimal effective dose every two weeks until discontinuation, or a hyperbolic tapering strategy, consisting of proportional dose reductions of approximately 20-25% every two weeks until discontinuation. Follow-up assessments will be conducted regularly over a 36-week period.

The primary outcome is the proportion of participants who fail to discontinue the antidepressant within the predefined tapering schedule (allowing a limited tolerance period) or who re-initiate antidepressant treatment during the 16 weeks following discontinuation. Secondary outcomes include measures of safety, tolerability, acceptability, clinical effectiveness, and cost-effectiveness, as well as withdrawal symptoms, relapse of depressive or anxiety symptoms, and adherence to the tapering schedule.

Participants and recruiting clinicians will not be blinded to treatment allocation, while outcome assessors and the biostatistician will remain blinded until completion of the study to minimize detection bias. The study aims to provide pragmatic evidence to inform clinical practice and guideline development regarding optimal strategies for antidepressant discontinuation.

DETAILED DESCRIPTION:
Antidepressants (ADs) are effective in the treatment of moderate-to-severe depression and anxiety disorders and are recommended by national and international clinical guidelines, although concerns about over-prescribing persist. In Italy, AD consumption increased by over 10% between 2014 and 2020. Selective serotonin reuptake inhibitors (SSRIs) account for approximately 70% of AD prescriptions and around half of total AD-related expenditure. Across most countries, AD prescribing has increased steadily, largely driven by use in general practice and by longer treatment duration.

For individuals experiencing a first depressive episode, evidence-based guidelines recommend continuing AD treatment for 6-9 months after clinical response. Meta-analytic evidence suggests a similar risk of relapse for maintenance periods ranging from six months to over one year. Treatment duration may vary according to illness severity and recurrence, with at least two years commonly recommended in cases of multiple episodes with functional impairment. In Italy, approximately one in three individuals continue AD treatment beyond 12 months, raising concerns about potentially inappropriate long-term or indefinite prescribing.

Prolonged AD use is associated with an increased risk of long-term adverse effects, including sexual dysfunction, weight gain, emotional blunting, and cardiovascular conditions. Discontinuation of ADs may also lead to withdrawal symptoms, which can be clinically relevant in a substantial proportion of patients. Several clinical factors appear to increase the risk of withdrawal, and it has been suggested that, for some individuals, disabling withdrawal symptoms rather than relapse may be the primary reason for unsuccessful discontinuation.

Randomized controlled trials indicate that discontinuing ADs is associated with a higher risk of relapse compared with continuation. However, discontinuation schedules used in many trials are rapid or abrupt, potentially increasing withdrawal symptoms that may be misclassified as relapse and thereby inflating relapse estimates. There is broad agreement that gradual tapering may reduce withdrawal symptoms, but most clinical guidelines provide only generic recommendations, often implying a linear dose reduction approach that remains standard in routine practice.

Alternative tapering strategies have been proposed, most notably hyperbolic tapering, which involves proportional dose reductions over longer periods. This approach is based on the nonlinear relationship between dose and receptor occupancy and may require tapering periods ranging from several months to over one year. Hyperbolic tapering often necessitates very low doses that are not readily achievable with standard marketed formulations, raising feasibility, regulatory, and policy challenges. To date, no randomized trials have directly compared different tapering strategies.

Against this background, there is a clear need for experimental evidence comparing hyperbolic and linear tapering approaches in routine clinical practice. The DISCARD study is a pragmatic, multicentre randomized trial designed to address this gap by comparing hyperbolic versus linear tapering in adults with currently remitted depressive disorders who have been taking ADs for at least six months and for whom discontinuation is clinically appropriate.

Participants will be recruited across four university psychiatric units in Italy, with methodological support provided by a fifth academic centre. General practitioners and other specialists will be involved in identifying potentially eligible individuals. After providing informed consent and completing baseline assessments, participants will be randomized to either a linear or a hyperbolic tapering strategy according to predefined schedules tailored to the starting dose. Follow-up assessments will be conducted regularly over a 36-week period using validated measures of depressive symptoms, anxiety symptoms, withdrawal symptoms, quality of life, and social functioning. Outcome assessors and the biostatistician will remain blinded to treatment allocation.

The primary outcome is the proportion of participants who fail to discontinue the AD within the predefined tapering schedule or who re-initiate AD treatment during the 16 weeks following discontinuation. Secondary outcomes include non-adherence to the tapering schedule, occurrence and severity of withdrawal symptoms, clinical relapse, early study discontinuation, and use of predefined rescue strategies. This study is designed to generate pragmatic evidence on the comparative effectiveness, feasibility, safety, and cost-effectiveness of hyperbolic versus linear tapering strategies in everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above;
* diagnosed with a depressive disorder, single episode (ICD-11, 6A70) or recurrent (ICD-11, 6A71);
* currently taking a selective serotonin reuptake inhibitor (SSRI), serotonin and norepinephrine reuptake inhibitor (SNRI), tricyclic antidepressant (TCA), or vortioxetine for the treatment of depression;
* the current AD has been taken for at least 6 months;
* the current AD has been on a stable dose over the last 2 months;
* a score ≤9 on the PHQ-9 and ≤5 on the GAD-7 at study enrolment;
* DSM-5-TR criteria for a depressive episode are not met at the time of recruitment;
* no clinical evidence of moderate-to-severe symptoms in the last 6 months, as assessed by the recruiting clinician;
* discontinuing the AD is clinically indicated by the recruiting clinician, and agreed to by the participant in a shared decision-making process;
* uncertainty about which discontinuation strategy would be best for the participant;
* the participant is willing to sign the informed consent to participate to the study.

Exclusion Criteria:

* comorbid schizophrenia-spectrum disorders, bipolar disorder, or dementia, as formally diagnosed by a psychiatrist, neurologist, geriatrician, or other specialists;
* current treatment with more than one AD at therapeutic doses;
* current treatment with ADs of other classes (e.g., mirtazapine, agomelatine, bupropion, for which the evidence on the risk of withdrawal is unclear), alone or in combination with other ADs;
* conditions or medications that contraindicate the use of any AD according to the Summary of Product Characteristics of included ADs (synthetically reported in Table 1) (e.g., current symptoms of mania);
* current treatment with benzodiazepines above the dose of 2.5 mg equivalents of lorazepam per day (corresponding to clonazepam 1.2 mg/day; alprazolam 1.2 mg/day; diazepam 19 mg/day);
* pregnancy or willingness to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Who Do Not Successfully Discontinue Antidepressant Treatment Within 16 Weeks | 16 weeks
  Proportion of participants who fail to successfully discontinue the antidepressant treatment, defined as either:
  1. continued use of the antidepressant beyond the predefined tapering schedule (allowing a tolerance period of up to 15% of the total tapering duration), or
  2. re-initiation of any antidepressant medication for any reason (e.g., withdrawal symptoms, recurrence of depressive or anxiety symptoms).

SECONDARY OUTCOMES:
Proportion of Participants Who Fail to Discontinue Antidepressant Treatment by the End of the Predefined Tapering Schedule | Up to the end of the predefined tapering period
  Proportion of participants who do not complete antidepressant discontinuation by the end of the predefined tapering schedule, regardless of reason
Proportion of Participants Who Re-initiate Antidepressant Treatment Within 16 Weeks After Discontinuation | Up to 16 weeks after complete antidepressant discontinuation
  Proportion of participants who restart any antidepressant medication for any reason after successful completion of the tapering schedule.
Proportion of Participants Non-adherent to the Predefined Antidepressant Tapering Schedule | Up to the end of the predefined tapering period
  Proportion of participants who deviate from the predefined tapering schedule for any reason.
Mean of DESS highest overall scores | Up to the end of the 16-weeks follow-up period
  A mean of the highest scores reached by each patient on the modified Discontinuation-Emergent Signs and Symptoms Scale (DESS)
Proportion of participants leaving the study early due to any reason without meeting criteria for the primary outcome | Up to the end of the 16-weeks follow-up period
  This includes people who do not attend follow-up visits and cannot be contacted, people who refuse to be involved in follow-up assessments, or people who die during the tapering or the follow-up for reasons unrelated to withdrawal symptoms or relapse.

OTHER OUTCOMES:
Proportion of participants requiring "rescue strategies" to address withdrawal symptoms | Up to the end of the 16-weeks follow-up period
  Proportion of participants requiring one or more "rescue strategies" (ie, benzodiazepines, gabapentinoids, or other mediacations) to address withdrawal symptoms during the tapering phase and the 16-weeks follow-up period
Time to clinical relapse | Up to the end of the 16-weeks follow-up period
  Time elapsed from randomization to clinical relapse, defined as having at least moderately severe depression or anxiety symptoms, namely a score ≥15 on the PHQ-9 or ≥10 on the GAD-7, up until the end of the 16-weeks follow-up period
Proportion of participants with "withdrawal-associated relapse" | Up to the end of the 16-weeks follow-up period
  Proportion of participants experiencing "withdrawal-associated relapse", defined as having a score ≥15 on the PHQ-9 or ≥10 on the GAD-7 within 4 weeks after the participant experienced "clinically relevant" withdrawal symptoms during the tapering phase and the 16-weeks follow-up period
PHQ-9 mean overall score | Up to the end of the 16-weeks follow-up period
  PHQ-9 mean overall score at the end of 16-weeks follow-up period
GAD-7 mean overall score | Up to the end of the 16-weeks follow-up period
  GAD-7 mean overall score at the end of 16-weeks follow-up period
Proportion of participants with suicidal behaviours | Up to the end of the 16-weeks follow-up period
  Proportion of participants with suicidal behaviours (including suicidal ideation, as reported by the participant, or according to a score ≥2 on the item 9 of the PHQ-9, suicide attempt, and deaths by suicide) at the end of 16-weeks follow-up period
Short Form 12 Health Survey (SF-12) Mental Component Summary mean score | Up to the end of the 16-weeks follow-up period
  Short Form 12 Health Survey (SF-12) mean score on the Mental Component Summary at the end of the 16-weeks follow-up period
Social Adaptation Self-evaluation Scale (SASS) mean score | Up to the end of the 16-weeks follow-up period
  Social Adaptation Self-evaluation Scale (SASS) mean score at the end of the 16-weeks follow-up period

IPD SHARING:
Plan to Share IPD: Yes
Once the dataset is completed, it will be uploaded to the online repository EUDAT-B2-SHARE, and will be made available after a motivated request, which will be discussed by the study's leading authors.
Supporting Information: Study Protocol, SAP, ICF